CLINICAL TRIAL: NCT04277975
Title: A Randomized Trial of Liberal vs. Restricted Post-discharge Opioid Prescribing Following Midurethral Sling
Brief Title: Liberal vs. Restricted Post-discharge Opioid Prescribing Following Midurethral Sling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jaime Long, Assistant Professor, Department of Obstetrics and Gynecology, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY13951
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Postoperative Pain; Opioid Use
Keywords: midurethral sling; opioid
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A: liberal post-discharge opioid prescribing (Active Comparator): Standardized postoperative instructions on non-opioid pain control + liberal opioid prescription provided prior to surgery (standard prescription for opioid prescribed prior to surgery)
  Interventions: Other: Restricted post-discharge opioid prescribing
- B: restricted post-discharge opioid prescribing (Experimental): Standardized postoperative instructions on non-opioid pain control + opioid prescribed only 'as needed' after discharge
  Interventions: Other: Liberal post-discharge opioid prescribing

INTERVENTIONS:
Other: Liberal post-discharge opioid prescribing — Opioid prescribed all patients opioids 'in case they are needed' prior to surgery
  Arms: B: restricted post-discharge opioid prescribing
Other: Restricted post-discharge opioid prescribing — Opioid only if needed after discharge
  Arms: A: liberal post-discharge opioid prescribing

SUMMARY:
The specific objective of this proposal is to evaluate pain and opioid use following a midurethral sling (MUS) under two different opioid prescribing schemes. The central hypothesis is that, in spite of the fact that opioids are often routinely prescribed by many surgeons following this procedure, most patients do not require them for pain control, and patients who are not prescribed postoperative will have similar pain scores and pain control satisfaction compared with patients who are routinely prescribed a standard amount of opioids for postoperative pain control.

DETAILED DESCRIPTION:
The investigators have 3 specific aims:

Specific Aim #1: Compare patients' postoperative pain experience and satisfaction with pain control using two different opioid prescribing schemes.

The investigators' working hypothesis is that postoperative pain control and satisfaction will be non-inferior between patients routinely prescribed opioids vs. those not routinely prescribed opioids prior to surgery.

Participants will be asked to complete a pain diary and assessment of their pain control satisfaction postoperatively. Pain control will be assessed by Likert scores (0-10) and satisfaction with pain control will be queried using an integer scale of 0-5 using REDCap or paper survey for the first 7 days postoperatively.

Specific Aim #2: Examine the opioid use of patients following midurethral sling.

The investigators will test the hypothesis that most patients who undergo MUS do not use prescribed opioid regardless of prescription scheme.

Given the investigators' standard of care preoperative education, including detailed instruction on non-opioid related pain management, they will prospectively examine the use of opioids after MUS under two different opioid prescribing routines. Women who agree to participation will be randomized to either be discharged home from surgery with a standard opioid prescription vs. only prescribed opioids if requested. The amount of opioid used will be collected via REDCap or paper survey for the first 7 days postoperatively. Investigators will also assess the subsequent requests for opioid prescription (among those not routinely given opioid prescription at discharge) or refill (among those who are initially given a standard amount of opioid upon discharge).

Specific Aim #3: Predict postoperative pain and opioid use after MUS with a brief psychometric questionnaire.

The investigators will leverage brief psychometric survey instruments in combination with individual demographic and clinical factors to predict postoperative pain and opioid use following MUS. They will seek to identify patients at risk for higher opioid needs or other pain interventions preoperatively, with a view to target education, prevention, and interventions on this population.

The project is original in comparing current clinical prescribing patterns with restrictive opioid prescribing. It capitalizes on providers' new ability to electronically prescribe opioids for patients who require them after discharge from the hospital, thereby decreasing the potential impact on patients and providers if prescribed opioid is requested once the patient has been discharged. The proposed work is innovative, because it examines recently developed psychometric survey instruments to identify patients at risk of postoperative pain. At the completion of this project, it is the investigators' expectation that the combination of work proposed in aims 1 -3 will optimize prescribing of opioids following this common MUS procedure, reducing the potential for both excessive opioid use (and adverse sequelae) postoperatively as well as unused opioid for subsequent misuse.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo isolated midurethral sling after evaluation and discussion with surgeon
* Consent to participate in this study

Exclusion Criteria:

* Pregnant or breast feeding
* Cognitively impaired women
* Pre-existing diagnosis of opioid use disorder
* Patients with chronic daily opioid use
* Prisoners
* Non-English speaking or inability to read, as a result of the need to read and report daily results in English
* Allergy to oral opioids used in this study (oxycodone)
* Significant contraindications (allergy, severe hepatic or renal compromise, or other medical conditions deemed by surgeon) to the use of both NSAIDs (ibuprofen, naproxen) and acetaminophen

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 84 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Pain score on postoperative day 1 | postoperative day 1
  Numeric score of pain at end of day (0-10 with 10 being the worst imaginable pain)

SECONDARY OUTCOMES:
Satisfaction with pain control | postoperative day 7 daily scores will be assessed
  scale of 1-5
The number of opioid pills used by those to whom they were prescribed | postoperative day 7 daily scores will be assessed
  Count of opioid pills used after surgery
Calls for new opioid prescriptions or refills postoperatively | postoperative day 7 daily outcome will be assessed
  Phone calls or office visits to obtain pain medication prescription
Psychometric survey and clinical/demographic factors associated with opioid use postoperatively | Upon enrollment
  Validated survey scores

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State College of Medicine, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] As-Sanie S, Till SR, Mowers EL, Lim CS, Skinner BD, Fritsch L, Tsodikov A, Dalton VK, Clauw DJ, Brummett CM. Opioid Prescribing Patterns, Patient Use, and Postoperative Pain After Hysterectomy for Benign Indications. Obstet Gynecol. 2017 Dec;130(6):1261-1268. doi: 10.1097/AOG.0000000000002344. PMID 29112660
- [Result] Howard R, Fry B, Gunaseelan V, Lee J, Waljee J, Brummett C, Campbell D Jr, Seese E, Englesbe M, Vu J. Association of Opioid Prescribing With Opioid Consumption After Surgery in Michigan. JAMA Surg. 2019 Jan 1;154(1):e184234. doi: 10.1001/jamasurg.2018.4234. Epub 2019 Jan 16. PMID 30422239
- [Result] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Result] Brummett CM, Waljee JF, Goesling J, Moser S, Lin P, Englesbe MJ, Bohnert ASB, Kheterpal S, Nallamothu BK. New Persistent Opioid Use After Minor and Major Surgical Procedures in US Adults. JAMA Surg. 2017 Jun 21;152(6):e170504. doi: 10.1001/jamasurg.2017.0504. Epub 2017 Jun 21. PMID 28403427
- [Result] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Result] Hill MV, McMahon ML, Stucke RS, Barth RJ Jr. Wide Variation and Excessive Dosage of Opioid Prescriptions for Common General Surgical Procedures. Ann Surg. 2017 Apr;265(4):709-714. doi: 10.1097/SLA.0000000000001993. PMID 27631771
- [Derived] Morgan BM, Long JB, Boyd SS, Davies MF, Kunselman AR, Stetter CM, Andreae MH. Liberal vs. restricted opioid prescribing following midurethral sling dataset. Data Brief. 2023 Apr 12;48:109144. doi: 10.1016/j.dib.2023.109144. eCollection 2023 Jun. PMID 37383763
- [Derived] Long JB, Morgan BM, Boyd SS, Davies MF, Kunselman AR, Stetter CM, Andreae MH. A randomized trial of standard vs restricted opioid prescribing following midurethral sling. Am J Obstet Gynecol. 2022 Aug;227(2):313.e1-313.e9. doi: 10.1016/j.ajog.2022.05.010. Epub 2022 May 10. PMID 35550371